CLINICAL TRIAL: NCT06049875
Title: Characteristics Associated With Duration of Home Hospitalization in Internal Department Versus Hospital in Internal Ward
Brief Title: Characteristics Associated With Duration of Home Hospitalization in Internal Department Versus Hospitalization in the Hospital in Internal Ward
Acronym: ARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Gad Segal, prof.Gad.Segal, Sheba Medical Center
Other Study IDs: Sheba 0096 GS 2023 CTIL
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Home Hospitalization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home Hospitalization: Patients who arrived at the emergency department and were discharged to home hospitalization or were hospitalized for a day and discharged to comprehensive home hospitalization under the management of a remote internist and a nurse who will make home visits on a daily basis.
- Internal Ward Hospitalization: Patients who arrived at the emergency department and received a regular treatment.

SUMMARY:
According to data from the OECD - Organization for Economic Co-operation and Development, the hospitalization crisis in Israel's hospitals is getting worse, both in relation to previous years in the State of Israel and in comparison to other countries [1]. There is an increase in life expectancy and the rate of aging of the population, which results in an increase in the number of beds in hospitals in relation to the growth rate of the population in need of treatment [2]. Furthermore, the government does not have the ability or an understandable plan for a significant and rapid increase in the number of hospital beds in the country. Instead, there is a recognition and a strategic decision by government officials in Israel, backed by the publication of relevant support tests [3], to develop hospitalization alternatives to hospital beds, primarily hospitalization within the community in the patient's natural environment, i.e. at home [4]. In a meta-analysis performed on patients with chronic diseases, it was found that the duration of treatment received by patients at home was 5.4 days longer compared to patients receiving treatment at the hospital, the risk of mortality was the same, re-hospitalization was lower among the patients hospitalized at home and the risk of worsening of the medical condition was smaller in 26 percent in hospitalization at home compared to hospitalization in the hospital [5]. For the patient receiving long-term care, it is extremely essential to be in a familiar and safe environment. Additional advantages to home hospitalization are a decrease in the chances of infection compared to the hospital and support from family members, both emotionally and physically [6].

Around the world, more and more experience is being accumulated in operating home hospitalizations as a substitute for hospitalization in a hospital. Comparative studies in diverse populations showed, already 20 years ago, that hospitalization at home is preferable to hospitalization in a hospital when it comes to the quality of life in a supportive and familiar environment [7]. However, the issue of the economic viability of home hospitalizations, whose cost was higher in the past, remains under question. There are studies that show a decrease in the cost of treatment in the home environment even in complex treatments and by professional teams [8]. Technological developments in the field of remote medicine have greatly contributed to improving the quality of care provided at home. Today, medical technology allows a patient who has been discharged from the hospital to be hospitalized at home, which allows the patient to continue to be treated at home through close medical and nursing supervision and advanced technological equipment. The technological development also allows cost reduction in different clinical settings such as: patients suffering from a flare-up of obstructive pulmonary disease [10,9], patients who are transferred to home hospitalization after surgery, elderly patients suffering from chronic diseases and needing hospitalization due to pneumonia and soft tissue infections, and patients suffering from exacerbation of heart failure [11]. The Ministry of Health and Welfare in the United States estimates that in 2030 one out of 5 Americans will be over the age of 65 and that home hospitalization is the preferred way to provide care to the patient as well as the optimal way in terms of costs [12]. This phenomenon will intensify the need for home hospitalization and will lead to improvements in the home sector [13].

At the Haim Sheba Tertiary Medical Center, they combine unique capabilities that make it particularly suitable for launching a home hospitalization service. The internal departments of the medical center are experienced in managing complex patients. The management of the departments is based on experts in internal medicine who have extensive experience in specializing in In the management of complex cases, with a high turnover of patients with mild and moderate degrees of severity, the hospital's position also matches the position of the relevant professional body - the Israeli Association of Internal Medicine - in regards to the launch of home hospitalization.

A center for innovation in digital health was established in Sheba, the purpose of which is to test and implement advanced technologies of remote medicine. Examining and operating these technologies, while having a unique collaboration with the companies that develop and manufacture them, places the innovation in an excellent opening position in terms of the ability to evaluate and operate the existing technologies in the hands of the doctors in the medical center.

DETAILED DESCRIPTION:
The purpose of the program:

Characterization, establishment and operation of a home hospitalization program managed by a hybrid division.

The target population is all patients who come from the community to the hospital's emergency room in Israel, who come to the emergency room for hybrid home hospitalization or hospitalization in an internal hospital department. The population accessible to the study is patients aged 18 and over who come to the emergency room for treatment and meet the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:Inclusion and exclusion criteria:

Criteria for the inclusion of the patients who come to the cognitive screening and who speak Hebrew to sign an informed consent with diagnoses:

* Respiratory infections in a patient who does not suffer from immunodeficiency
* Infection of the urinary tract in a patient who does not suffer from immunodeficiency

  * Soft tissue infection of the lower limbs in a patient who does not suffer from immunodeficiency
* Flare-up of chronic obstructive pulmonary disease in a patient who does not demonstrate respiratory failure in the emergency department
* Infection of the upper/lower digestive tract in a patient who does not suffer from immunodeficiency
* Starting the investigation of a prolonged febrile illness of unknown origin in a patient who does not suffer from immunodeficiency
* Flare-up of heart failure in a respiratory and hemodynamically stable patient - including hypoxemia

Exclusion Criteria:• Patients who are not cognitively fit

* Patients who do not speak Hebrew
* Patients who came to the emergency department with delirium
* Patients who do not have the appropriate conditions for home hospitalization - terminally ill, lack of family support, and lack of ability to operate technologies in a home setting
* Patients with hemodynamic, respiratory or neurological instability.
* Patients whose treatment requires the use of measures or drugs that cannot be provided in a hospital setting
* Unbalanced psychiatric patients
* Patients who live within a radius of more than 50 km from Sheba Hospital (according to the procedure of the Ministry of Health)
* Patients who are not interested in home hospitalization / or who were hospitalized during home hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — MALE&FEMAEL
Study Population: The target population is all patients who come from the community to the hospital's emergency room in Israel, who come to the emergency room for hybrid home hospitalization or hospitalization in an internal hospital department. The population accessible to the study is patients aged 18 and over who come to the emergency room for treatment and meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The length of hospitalization will differ between hospitalization in an internal ward and hospitalization at home. | 01/07/2023-01/12/2024
  We expect that the duration of home hospitalization will be shorter than that of hospitalization in an internal ward. This outcome will be measured using descriptive analysis.
The number of re-hospitalizations will differ between hospitalization in an internal ward and hospitalization at home. | 01/07/2023-01/12/2024
  We expect that the number of re-hospitalizations of home hospitalization will be lower than that of hospitalization in an internal ward. This outcome will be measured using descriptive analysis.
The level of satisfaction will differ between hospitalization in an internal ward and hospitalization at home. | 01/07/2023-01/12/2024
  We expect that the level of satisfaction of home hospitalization will be higher than that of hospitalization in an internal ward. This outcome will be measured using the PPEQ-15 questionnaire.
The cost of hospitalization will differ between hospitalization in an internal ward and hospitalization at home. | 01/07/2023-01/12/2024
  We expect that the cost of home hospitalization will be lower than that of hospitalization in an internal ward. This outcome will be measured using descriptive analysis.
Clinical outcomes will differ between hospitalization in an internal ward and hospitalization at home. | 01/07/2023-01/12/2024
  We anticipate differences in aspects of clinical deterioration of the patient, falls, new infection, delirium and death. This outcome will be measured using the NEWS-2 questionnaire.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Difference between tow independent mean -tow groups, Ramat Gan
  - Sheba Medical Center, Ramat Gan
  - Daniella Daliyot, Ramat Gan